CLINICAL TRIAL: NCT02563561
Title: A Multicenter, Multi-Arm, Randomized, Multi-Dose, Placebo-Controlled, Double-Blind, Phase 3 Study of Intravesical Apaziquone (EOquin®) as a Surgical Adjuvant in the Immediate Postoperative Period in Patients Undergoing Transurethral Resection for Non- Muscle Invasive Bladder Cancer
Brief Title: A Study of Intravesical Apaziquone as a Surgical Adjuvant in Participant Undergoing Transurethral Resection Bladder Tumor (TURBT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPI-EOQ-13-305
Record Dates: First submitted 2015-09-21; First posted 2015-09-30 (Estimated); Results first posted 2021-09-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Non-muscle invasive bladder cancer; Apaziquone; TURBT; Stage Ta, G1-G2
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Dose Apaziquone (Experimental): Participants were randomized to receive first dose of 4 mg of apaziquone by intravesical administration into the bladder at 60 ± 30 minutes post transurethral resection of bladder tumor (TURBT) on Day 1 via an indwelling 100% Silicone Foley catheter. Followed by second dose of placebo by intravesical administration via an indwelling catheter on Day 15 (±5 days).
  Interventions: Drug: Apaziquone; Other: Placebo
- 2 Dose Apaziquone (Experimental): Participants were randomized to receive first dose of 4 mg of apaziquone by intravesical administration into the bladder at 60 ± 30 minutes post TURBT on Day 1 via an indwelling 100% Silicone Foley catheter. Followed by second dose of 4 mg of apaziquone by intravesical administration via an indwelling catheter on Day 15 (±5 days).
  Interventions: Drug: Apaziquone
- Placebo (Placebo Comparator): Participants were randomized to receive first dose of matching placebo by intravesical administration into the bladder at 60 ± 30 minutes post TURBT on Day 1 via an indwelling 100% Silicone Foley catheter. Followed by second dose of matching placebo by intravesical administration via an indwelling catheter on Day 15 (±5 days).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apaziquone — One dose of apaziquone administered by intravesical administration
  Other Names: EOquin
  Arms: 1 Dose Apaziquone; 2 Dose Apaziquone
Other: Placebo — Matching placebo (containing 12 mg FD&C red #40, 15 mg sodium chloride, and 10 mg mannitol was supplied in identical appearing vials) by intravesical administration.
  Arms: 1 Dose Apaziquone; Placebo

SUMMARY:
This is a Phase 3, randomized, multicenter, multi-arm, placebo-controlled, double-blind study of apaziquone in participants with ≤4 non-muscle invasive bladder cancer (NMIBC), ≤3.5 centimeters (cm) in diameter, all of which must had been fully resected at TURBT.

In addition to Screening, participants underwent an assessment of urothelial carcinoma of the bladder via cystoscopy for clinically apparent tumor Ta, G1-G2.

Following TURBT on Day 1, eligible participants were randomized to one of three treatment arms in a 1:1:1 ratio.

Arm 1 : One dose of Apaziquone. Arm 2 : Two Doses of Apaziquone. Arm 3 : Placebo. Primary endpoint was to evaluate the Time to Recurrence with either a one instillation of 4 mg apaziquone or two instillations of 4 milligram (mg) apaziquone relative to placebo instillation following TURBT in a participant with NMIBC who received TURBT.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, multicenter, multi-arm, placebo-controlled, double-blind study of apaziquone in participants with ≤4 non-muscle invasive bladder tumors, ≤3.5 cm in diameter, all of which must have been fully resected at TURBT.

In addition to Screening, participants underwent an assessment of urothelial carcinoma of the bladder via cystoscopy for clinically apparent tumor Ta, G1-G2.

Following TURBT on Day 1, eligible participants were randomized to one of three treatment arms in a 1:1:1 ratio :

Arm 1 : One Dose of Apaziquone:

* Day 1: administration of 4 mg of apaziquone 60±30 minutes post-TURBT
* Day 15 (±5 days): administration of placebo

Arm 2 : Two Doses of Apaziquone :

* Day 1: administration of 4 mg of apaziquone 60±30 minutes post-TURBT
* Day 15 (±5 days): administration of 4 mg of apaziquone

Arm 3: Placebo :

* Day 1 : administration of placebo 60±30 minutes post-TURBT
* Day 15 (±5 days) : administration of placebo

Once randomized, Day 1 study drug instillation occurred 60 ±30 minutes post TURBT. Participants returned on Day 15 (±5 days) for a second instillation unless their pathology results showed non Ta, G1-G2 histology; in the absence of local pathology results by the Day 15 visit, participants received a second instillation of study drug. All histology specimens were reviewed by a local pathology laboratory and all clinical treatment decisions and study analyses were based on the local pathology review. Participants whose pathology was other than Ta, G1-G2 were followed for safety at Day 35 (±5 days) from the last dose of study drug and then discontinued from the study.

Participants with pathology confirmed Ta, G1-G2 disease were followed according to the schedule below :

* Cystoscopic examination and urine cytology every 90 days (±10 days) (calculated from date of TURBT) through 24 months for tumor recurrence and progression.
* If at any time during the 24 months follow up period there was a tumor recurrence, the participant continued on study with follow-up cystoscopic examination and urine cytology every 90 days (±10 days) (calculated from date of TURBT) through the end of 24 months. Participants with a recurrence were permitted to have a follow-up TURBT.
* If at any time during the 24 months follow up period there was a tumor recurrence and/or participant started on another therapy, the participant was followed by telephone, for safety every 90 days (±10 days) (calculated from date of TURBT) through the end of 24 months.

Duration of Study: The duration of the study for each participant was approximately 24 months including:

* Screening Period : 30-days
* Treatment Period : Day 1 and Day 15 (±5 days)
* Safety and Follow-up Period: 24-months

ELIGIBILITY:
1. Participant must have had a diagnosis with urothelial carcinoma of the bladder with clinically apparent tumor Ta, G1-G2.
2. Participant had ≤4 tumors, none of which exceeded 3.5 cm in diameter.
3. Participant must have been willing to give written informed consent, able to adhere to dosing and visit schedules, and meet all study requirements.
4. Participant was at least 18 years of age at randomization.
5. Participant must have been willing to practice two forms of contraception, one of which must have been a barrier method, from study entry until at least 35 days after the last dose of the study drug.
6. Female participant of childbearing potential must have had a negative pregnancy test within 30 days prior to randomization. Female participant who was postmenopausal for at least 1 year (defined as more than 12 months since last menses) or were surgically sterilized did not require this test.

Exclusion Criteria:

1. Participant had an active concurrent malignancy/life-threatening disease. If there was a history of prior malignancies/life-threatening diseases, the participant was to be disease-free for at least 5 years. Participant with other prior malignancies less than 5 years before study entry could have still been enrolled if they had received treatment resulting in complete resolution of the cancer and currently had no clinical, radiologic, or laboratory evidence of active or recurrent disease.
2. Participant had positive urine cytology for malignancy at Screening.
3. Participant had an active uncontrolled infection, including a urinary tract infection, underlying medical condition, or other serious illness that would impair the ability of the participant to receive protocol treatment.
4. Participant had used any investigational drugs, biologics, or devices within 30 days prior to study treatment or planned to use any of these during the course of the study.
5. Participant had any prior intravesical chemotherapy, immunotherapy, or previous exposure to apaziquone.
6. Participant had or has ever had

   * Upper tract Transitional Cell Carcinoma (TCC).
   * Urethral tumor (prostatic urethra included).
   * Any invasive bladder tumor known to be other than tumor Ta, G1-G2.
   * Any evidence of lymph node or distant metastasis.
   * Any bladder tumor with histology other than TCC.
   * Carcinoma in situ (CIS).
7. Participant had a tumor in a bladder diverticulum.
8. Participant had received any pelvic radiotherapy (including external beam and/or brachytherapy.)
9. Participant had a bleeding disorder or a screening platelet count <100×10^9/L.
10. Participant had screening hemoglobin <10 milligrams per deciliter (mg/dL).
11. Participant had any unstable medical condition that would make it unsafe to undergo TURBT.
12. Participant had a history of interstitial cystitis.
13. Participant had a history of allergy to red color food dye.
14. For a participant with a recurrent tumor, the participant had at least a 6-month cystoscopically-confirmed tumor-free interval between the last tumor recurrence and screening cystoscopic examination.
15. Participant was pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Urology Center of Colorado, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who underwent Transurethral Resection for Non-Muscle Invasive Bladder Cancer (NIMBC) were enrolled at 17 investigative sites in the United States and Canada from 09 Oct 2015 to 10 March 2017.
Pre-assignment Details: A total of 62 participants were randomized into the study, out of which 6 participants completed the study.
Period: Overall Study
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
Started | 19 | 23 | 20
Safety Population | 19 | 21 | 17
Completed | 1 | 2 | 3
Not Completed | 18 | 21 | 17
Not completed — Histology Other than Ta, G1-G2 | 3 | 6 | 6
Not completed — Withdrew of Consent | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Participant Had Recurrence and Received Therapy | 4 | 2 | 1
Not completed — Investigator Decision | 3 | 4 | 2
Not completed — Sponsor Decision | 5 | 2 | 4
Not completed — Other | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants classified according to the actual treatment received, regardless of random assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 17 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.2) | 66.6 (12.4) | 66.1 (12.4) | 66.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 18
  Male | 14 | 14 | 11 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 18 | 21 | 14 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 18 | 20 | 17 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence
Description: Time from randomization to the date of histologically confirmed recurrence of bladder cancer. A recurrence was defined as any pathologically confirmed disease of ≥Ta tumor histology or carcinoma in situ (CIS) post-treatment.
Time Frame: From randomization to the date of first histologically confirmed recurrence of bladder cancer (up to 1.5 years)
Population: Data for this outcome measure was not collected due to early termination of study.
Groups:
- 1 Dose Apaziquone: Participants were randomized to receive first dose of 4 mg of apaziquone by intravesical administration into the bladder at 60 ± 30 minutes post TURBT on Day 1 via an indwelling 100% Silicone Foley catheter. Followed by second dose of placebo by intravesical administration via an indwelling catheter on Day 15 (±5 days).
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: 2-Year Recurrence Rate
Description: The percentage of participants with histologically confirmed recurrence of the bladder tumor at any time after randomization and on or before Year 2. A recurrence was defined as any pathologically confirmed disease of ≥Ta tumor histology or CIS post-treatment.
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: 1-Year Recurrence Rate
Description: The percentage of participants with histologically confirmed recurrence of the bladder tumor at any time after randomization and on or before Year 1. A recurrence was defined as any pathologically confirmed disease of ≥Ta tumor histology or CIS post-treatment.
Time Frame: 1 year
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time to Progression
Description: Time to disease progression was defined as the time from randomization to the first disease progression. The development of T2 or greater disease was only included in the assessment of time to disease progression.
Time Frame: From randomization to the date of first disease progression (up to 1.5 years)
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Adverse Events, Serious Adverse Events (SAEs), TEAEs Leading to Discontinuation and Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it did not necessarily have to have a causal relationship with this treatment. TEAEs were adverse events that occurred from the first dose of study treatment until 40 days after the last dose of study drug administration or 40 days after the date of participant early discontinuation. Treatment-related AEs included TEAEs with relationship to study treatment reported as possible, probable, definite, or missing. An SAE was an AE resulting in any of the outcomes: death; initial/prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 1.5 Years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
Number analyzed (Participants) | 19 | 21 | 17
Participants
  TEAEs | 10 | 13 | 7
  Treatment-Related AEs | 4 | 4 | 5
  SAEs | 0 | 2 | 1
  TEAEs Leading to Discontinuation | 0 | 0 | 0
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1.5 years
Description: Safety Population included all randomized participants classified according to the actual treatment received, regardless of random assignment.
Arm/Group | 1 Dose Apaziquone | 2 Dose Apaziquone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/21 | 1/17
Other Adverse Events (participants affected / at risk) | 10/19 | 12/21 | 7/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Dose Apaziquone (N=19) | 2 Dose Apaziquone (N=21) | Placebo (N=17)
Bladder Perforation (Renal and urinary disorders) | 0 | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Dose Apaziquone (N=19) | 2 Dose Apaziquone (N=21) | Placebo (N=17)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Adrenal Mass (Endocrine disorders) | 1 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cervical Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Bladder Pain (Renal and urinary disorders) | 2 | 2 | 0
Bladder Spasm (Renal and urinary disorders) | 2 | 4 | 0
Dysuria (Renal and urinary disorders) | 4 | 7 | 2
Haematuria (Renal and urinary disorders) | 1 | 3 | 1
Micturition Urgency (Renal and urinary disorders) | 2 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 2 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary Hesitation (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 1 | 0
Urine Abnormality (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated as per Sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT02563561/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT02563561/SAP_001.pdf